CLINICAL TRIAL: NCT03544450
Title: Effectiveness of Non-medical Health Worker (NMHW) Led Counseling on Common Mental Disorders in Rural Mid-western Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Victims of Torture, Nepal (Other)
Collaborators: Physicians for Social Responsibility, Finland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CounselingCvict
Record Dates: First submitted 2016-04-25; First posted 2018-06-01 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Mental Disorders; Psychological Distress; Depression; Anxiety; Coping
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychosocial counselling + Enhanced usual care (EUC) (Experimental): This arm receives psychosocial counselling from the counsellor as well as enhanced usual care from health worker
  Interventions: Behavioral: Psychosocial counselling; Other: Enhanced Usual Care
- Enhanced Usual Care (EUC) (Active Comparator): This arm receives enhanced usual care from health worker
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Psychosocial counselling — Individuals with psychological distress receive psychosocial counselling and enhanced usual care. The psychosocial the counselling process consists of: (i) introduction, explanation and rapport building; (ii) assessment of and understanding of the problem (including looking for positive assets); (iii) goal setting (asking the client what outcomes are preferred); (iv) problem management (exploring and identifying solutions, brainstorming, working with existing coping strategies, using social and cultural resources, and additional techniques such as relaxation and psycho-education); (v) implementation (making a plan of action and transition); and, finally, (vi) termination of counselling (including closing and follow-up)." Enhanced usual care is provided by health workers, who have already been trained on diagnosis and treatment of common mental disorders, and usage of basic psychosocial counseling skills (communication, listening and basic emotional support).
  Arms: Psychosocial counselling + Enhanced usual care (EUC)
Other: Enhanced Usual Care — Enhanced usual care is provided by health workers, who have already been trained on diagnosis and treatment of common mental disorders, and usage of basic psychosocial counseling skills (communication, listening and basic emotional support).

SUMMARY:
Psychological treatments may be provided by non-medical health workers (NMHW) to increase accessibility. Task shifting of screening and treatment of non-communicable diseases to non-medical health workers is both effective and cost-effective. A recent review included five randomized controlled trials to assess effectiveness of NMHW provided psychological interventions to treat common mental disorders and depression, and all five trials found the intervention beneficial over usual treatment.

The aim of this study is to assess the effectiveness of psychosocial counselling as practiced by non-medical psychosocial counsellors in improving the outcomes of persons with common mental disorders in a primary health care setting.

Patients with psychosocial distress will be randomized to receive either counseling + enhanced usual care or enhanced usual care by health workers. The hypothesis is that adding psychosocial counselling to enhanced usual care, will be more effective than enhanced care alone in reducing the symptoms of depression, anxiety and posttraumatic stress disorder and in improving day-to-day functioning of clients receiving services in primary health care settings.

If proven effective, non-medical health worker led counseling could be an affordable treatment to alleviate psychological suffering and improve functional capacity of Nepalese people.

DETAILED DESCRIPTION:
Statement of problem

Psychosocial interventions, such as counselling, are effective in improving social functioning in common mental disorders. Specifically, culturally adapted psychological treatments are effective in the treatment of depression, according to a recent meta-analysis.

Psychological treatments may be provided by non-medical health workers (NMHW) to increase accessibility. Task-shifting of screening and treatment of non-communicable diseases to non-medical health workers is both effective and cost-effective. A recent review included five randomized controlled trials to assess effectiveness of NMHW provided psychological interventions to treat common mental disorders and depression, and all five trials found the intervention beneficial over usual treatment.

In the MANAS trial in India, for example, those receiving the intervention were 55% more likely to recover from common mental disorders than the control group in public health facilities. The stepped-care intervention was provided by NMHWs who had received a two-month training in counselling. In Pakistan, a psychological treatment delivered by Lady Health Workers (NMHWs) resulted in 78% reduction in maternal depression, compared with usual care.

In Nepal, the need for psychosocial interventions led by NMHWs is high because of the very limited number of mental health professionals. Centre for Victims of Torture (CVICT) has extensive experience in developing psychosocial counseling services and training counsellors. CVICT has experienced that even a short intervention, including only 1-5 counselling sessions, leads to decreased mental distress. Positive feedback has been given both by the patients and the people working in primary health care. However, no rigorous research has been conducted on the effectiveness of counselling on the symptoms of common mental disorders. This will be the first study comparing the effectiveness of psychosocial counseling and enhanced usual care to enhanced usual in rural Nepal.

Conceptual framework

This trial will examine the added value of psychosocial counseling in individuals with psychological distress when provided together with enhanced usual care in rural health posts.

The psychosocial approach emphasizes the close connection between psychological aspects of an individual's experience (namely, thoughts, feelings and beliefs) and the wider social experience (namely, relationships with family, community and friends) as well as the broader social environment (i.e. culture, traditions, religion, socio-political environment). There is a dynamic relationship between the psychological and social effects of experiences on the individual person, with each continually influencing the other.

Psychosocial counselling starts with the complaints that a client brings into the session, and is aimed at decreasing disability. The client is assisted in dealing with problems himself/herself within a counselling process, or is sometimes referred to other existing resources if the counsellor feels that to be more appropriate. Specifically, the counselling process consists of: (i) introduction, explanation and rapport building; (ii) assessment of and understanding of the problem (including looking for positive assets); (iii) goal setting (asking the client what outcomes are preferred); (iv) problem management (exploring and identifying solutions, brainstorming, working with existing coping strategies, using social and cultural resources, and additional techniques such as relaxation and psycho-education); (v) implementation (making a plan of action and transition); and, finally, (vi) termination of counselling (including closing and follow-up). This process helps to reduce psychological distress experienced by the patients and is practiced by trained psychosocial counselors.

Enhanced usual care is provided by health workers, who have already been trained on diagnosis and treatment of common mental disorders, and usage of basic psychosocial counseling skills (communication, listening and basic emotional support).

It is important to note that in this conceptual framework psychosocial counselling is just one part of the spectrum of psychosocial care and dealing with distress in Nepal's context where there are other issues such as poverty, human rights abuses, gender based violence etc.

General objective

To assess the effectiveness of psychosocial counseling as practiced by non-medical psychosocial counselors in improve the outcomes of persons with common health disorders in primary health care setting.

Specific objective

To assess the effectiveness of psychosocial counselling on:

* reducing symptoms of depression and anxiety
* improving functional capacity
* improving coping and use of available resources

To assess acceptability of psychosocial counseling.

Study variables

Depressive symptoms, anxiety symptoms, coping mechanisms and usage of available resources, functional capacity

Covariates: Demographic variable (gender, age, socioeconomic position)

Study population

Residents of Dang

Study units

Individuals

Sampling methods

As this is a randomized controlled trial, randomization will be done using a randomization table. Participants coming to the health post for treatment of symptoms of psychological distress will be potential participants for this research. Individuals referred by the counselors during their field mental health promotion work will also be potential participants for this research. Individuals will be screened with the General Health Questionnaire (GHQ-12, validated Nepali version, and those who score 6 or more on will be invited to participate in the study. The Research Assistant will use the GHQ. In the Nepali context, score of 6 or more in the GHQ-12 reveals psychological distress. The GHQ-12 was validated using Likert scale in Nepal. Randomization will be done by a health worker at the health post. Research Assistant will be blinded to the study.

Sampling size

A sample size of 132 in each group will be required to detect a clinically important difference of three points on the Beck scale of depression (BDI: Beck Depression Inventory), using a two-tailed test of the difference between means and a power of 80%, and a significance level of 5%. Based on a previous study, we assume a standard deviation of 8.7 for BDI and also the calculation is based on the assumption that the measurements on BDI are normally distributed. However, considering the possible 30% dropout rates, we will need to recruit 176 individuals per group, 352 in total.

Data collection technique

Data will be collected on paper and stored safely in lockers. No names will appear on study forms. All participants will be read out consent forms and asked to sign on the form. All questions of the data tools will be read aloud and participants will be asked to choose which level they agree with on Likert's scale. RA's data and counselors data will be kept separately. Study coordinator will enter data into SPSS bi-weekly. Participants will be referred by the project counselors, female community health volunteers and health workers of other health posts to the centres for study/ treatment.

Data collection tools

For the Quantitative study, questionnaires will be used to collect the data from each group. The questionnaire will have five sections. The sections are: Socio and Demographic information, Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), World Health Organization Disability Assessment Schedule-II (WHODAS-II) and Resource and Coping Mechanism will be used. All in all tools are validated in Nepal and study area (Dang), availed in Nepali language and used by CVICT in their previous Research.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16
* GHQ-12 ≥ 6
* Willing to participate in the intervention and research program
* Able to communicate fluently in Nepali and to participate the required visits
* Resident in Dang for the subsequent 10 months

Exclusion Criteria:

* Age < 16
* GHQ-12 < 6
* Signs of severe mental health problems (i.e., psychotic features)
* Severe illnesses or conditions requiring immediate attentions( i.e., suicidal)
* Not willing to participate in the intervention and research program

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who have a response to treatment when assessed by change in the symptoms of depressive symptoms measured by Beck Depression Inventory | 0 months, 1 month, 6 months
  The range of scale is 0-63 scores and higher scores indicate higher levels of depression. Reduction of 50% or more from initial BDI score indicates response. The instrument is used at baseline, 1 month and 6 months in both groups.

SECONDARY OUTCOMES:
Change in the symptoms of anxiety assessed by Beck Anxiety Inventory | 0 months, 1 month, 6 months
  The range of scale is 0-63 scores and higher scores indicate higher levels of anxiety. The instrument is used at baseline, 1 month and 6 months in both groups.
Change in the functional capacity assessed by World Health Organisation Disability Assessment Schedule - II | 0 months, 1 month, 6 months
  The validated Nepali version of WHODAS-II includes 13 questions and the range of scale is 13-65 scores. Higher scores indicate lower level of functional capacity. The instrument is used at baseline, 1 month and 6 months in both groups.
Change in the symptoms of depression assessed by Beck Depression Inventory | 0 months, 1 month, 6 months
  The range of scale is 0-63 scores and higher scores indicate higher levels of depression. The instrument is used at baseline, 1 month and 6 months in both groups.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patel V, Weiss HA, Chowdhary N, Naik S, Pednekar S, Chatterjee S, De Silva MJ, Bhat B, Araya R, King M, Simon G, Verdeli H, Kirkwood BR. Effectiveness of an intervention led by lay health counsellors for depressive and anxiety disorders in primary care in Goa, India (MANAS): a cluster randomised controlled trial. Lancet. 2010 Dec 18;376(9758):2086-95. doi: 10.1016/S0140-6736(10)61508-5. Epub 2010 Dec 13. PMID 21159375
- [Background] Tol WA, Jordans MJ, Regmi S, Sharma B. Cultural challenges to psychosocial counselling in Nepal. Transcult Psychiatry. 2005 Jun;42(2):317-33. doi: 10.1177/1363461505052670. PMID 16114588